CLINICAL TRIAL: NCT04628195
Title: Cardiac Performance in Mechanically Ventilated Patients With Severe Pneumonia by SARS-CoV-2: Echo-COVID Study
Brief Title: Cardiac Performance in Mechanically Ventilated COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Clinica Alemana de Santiago (Other); Hospital Barros Luco Trudeau (Other); University of Chile (Other)
Responsible Party: Principal Investigator, Emilio Valenzuela, M.D. Intensivist, Pontificia Universidad Catolica de Chile
Other Study IDs: 200422002
Record Dates: First submitted 2020-11-10; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Acute Cor Pulmonale; Cardiac Failure
Keywords: Critical Care Echocardiography; Cardiac Function; Acute Cor Pulmonale; COVID-19; Mechanical Ventilation; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although COVID-19 affects primarily the respiratory system, several studies have shown evidence of cardiovascular alterations. Increased troponin levels were observed in a significant proportion of patients and this alteration was associated with higher mortality. In addition, case reports of cardiogenic shock or fulminant myocarditis have been communicated. Likewise, pulmonary embolism (PE), right ventricle dilation, and acute cor pulmonale (ACP) have also been described. Therefore, investigating cardiac function in COVID-19 is highly relevant, particularly in critically ill patients who are usually under sedation and mechanical ventilation, which may further impair cardiovascular function. Thus the objective is to determine the prevalence of left ventricle dysfunction and acute cor pulmonale, and its association with respiratory mechanics, in 100 consecutive critically ill COVID-19 patients, who were assessed with critical care echocardiography (CCE) within the first 24 hours of mechanical ventilation.

DETAILED DESCRIPTION:
The objective is to determine the prevalence of left ventricle dysfunction and acute cor pulmonale, and its association with respiratory mechanics, in 100 consecutive critically ill COVID-19 patients, who were assessed with critical care echocardiography (CCE) within the first 24 hours of mechanical ventilation.

Material and Methods This prospective, multicenter study was conducted between April and June 2020 in the intensive care unit (ICU) of four university-affiliated hospitals of Santiago, Chile. Local ethics committee of each center approved the study and waived the need to provide written informed consent (protocol ID: 200422002). All participating centers have expertise in CCE on clinical grounds.

The study population Were included systematically all consecutive patients with severe SARS-CoV-2 pneumonia, defined as respiratory failure requiring invasive mechanical ventilation (MV). Patients were included within the first 24 hours of MV. COVID-19 was confirmed by a positive polymerase chain reaction test. The main exclusion criteria were age under 18 years old, severe valvulopathy, poor ultrasound window and do-not-resuscitate status.

Demographic data, Acute Physiology and Chronic Health Evaluation II (APACHE), Sequential Organ Failure Assessment (SOFA) and respiratory system mechanics were recorded.

Echocardiography Transthoracic echocardiography was performed by intensivists trained in echocardiography in according to CCE. Echocardiographic measurements were obtained with a Vivid i echocardiography system (GE Medical Systems, Milwaukee, WI, USA), Philips CX 50 (Philips Healthcare, DA Best, The Netherlands), and Mindray M9 (Bio-Medical Electronics Co., Shenzhen, Chine), as used in each center. All patients were adapted to MV on continuous IV sedation during the echocardiographic assessment. Measurements were acquired at end-expiration and averaged over three consecutive cardiac cycles in according to current recommendations.

Standard echocardiographic views were acquired. Left ventricular systolic function was assessed by the left ventricular ejection fraction (LVEF), as measured with Simpson's modified rule. Based on LVEF patients were categorized in hyperkinetic (LVEF >60%), normokinetic (LVEF between 45% and 60%) and hypokinetic (LVEF <45%).

Cardiac output (CO) was calculated from the left ventricular outflow tract (LVOT) as described by Mclean et al. The diameter of the LVOT was taken from the long parasternal view. Pulsed wave Doppler samples were obtained at the LVOT from the apical view. Doppler velocity curves were manually traced and an average of three measures of velocity time integral (VTI) was calculated. The stroke volume (SV) was calculated as the product of the LVOT area and the VTI. The CO was calculated as the product of the SV and the heart rate obtained during measurement of the aortic VTI. Mitral annular plane systolic excursion (MAPSE) was obtained through an M-mode vector at the level of the mitral annulus at the LV lateral wall. MAPSE was measured in millimeters as described (5). Peak mitral annular myocardial velocity wave (s') was recorded at the level of the mitral annulus at the LV lateral wall with Tissue Doppler Imaging (TDI) as previously described.

Left ventricular diastolic function was assessed by mitral inflow pulsed wave Doppler, to measure early peak velocity (E) and atrial velocity (A). The early diastolic peak velocity (e') of the lateral mitral annulus was also measured with TDI. From these variables E/A and E/e' ratios were calculated. Diastolic function was categorized as normal, grade I to grade III according to current recommendations.

The presence of acute cor pulmonale was assessed through the relation between left and right ventricular end-diastolic areas (LVEDA and RVEDA), and by the presence of paradoxical septum motion. LVEDA and RVEDA were measured from the apical four chambers view, and the RVEDA/LVEDA ratio was calculated. Right ventricle (RV) dilatation was defined as RVEDA/LVEDA ratio > 0.6, ACP was defined as a dilated RV associated with the presence of paradoxical septum motion. Severe ACP was defined as a severely dilated RV (RVEDA/LVEDA ratio >1). Paradoxical septum motion was defined as end-systolic bulging of the interventricular septum toward the left ventricle, while analyzing loops in slow motion. It indirectly assesses RV performance and RV end-diastolic pressures. The paradoxical septum motion was assessed on the four-chamber view. In addition, RV systolic function was assessed by the tricuspid annular plane systolic excursion (TAPSE) obtained through an M-mode vector at the level of the tricuspid annulus.

Hemodynamic assessment The hemodynamic profile was based on cardiac index (CI), patients were categorized as hypodynamic (CI<2 L⋅min-1⋅m2), normodynamic (CI between 2 and 4 L⋅min-1⋅m2) and hyperdynamic (CI>4 L⋅min-1⋅m2). Hemodynamic variables and norepinephrine doses were recorded. Maximum and minimum inferior vena cava (IVC) diameter was measured in M-mode tracing from a longitudinal subcostal view. Fluid responsiveness was assessed by either the respiratory variations of inferior vena cava (IVC), or by the arterial pulse pressure variation (PPV).

The PiCCO (Continuous Cardiac Output Pulse Index) device was used in thirty patients to assess cardiac output (CO). An average of three consecutive thermodilution measurements was used. Other variables such as global end-diastolic index (GEDI), intrathoracic blood volume index (ITBVI), systemic vascular resistance index (SVRi), cardiac function index (CFi), global ejection fraction (GEF), extravascular lung water index (ELWI), and pulmonary vascular permeability index (PVPI), were recorded.

Tissue perfusion was assessed by capillary refill time (CRT) and lactate levels. The peripheral perfusion index (PFI) derived from the photoelectric plethysmography signal of pulse oximetry was also used.

Computer tomography (CT) pulmonary angiography was performed based on the clinical suspicion of PE.

Biomarkers High-sensitive Troponin T and D-Dimer (DD) concentrations were measured simultaneously with echocardiographic assessment. Increases in Troponin T were defined as a value >14ng/l.

Statistical Analysis As the study was descriptive sample size but was arbitrarily set at 100 consecutive patients. Normality was tested by Kolmogorov-Smirnov test. The continuous data is presented as mean ± standard deviation or as median and interquartile ranges, depending on the distribution. Comparisons between groups were analyzed by t-test or Wilcoxon rank-sum (WRS) test according to data distribution. Percentages were analyzed using two-proportion z-test. Categorical variables were compared with chi square test. Pearson or Spearman correlation was performed according to data distribution.

In order to identify independent predictors for mortality, a multivariate regression analysis was carried out including all variables of interest associated with mortality in a univariate analysis (p value < 0.05) and adjusting for the other covariates of the logistic regression model. The discrimination of the model was assessed by the area under the receiver operating characteristic (ROC) curve. Statistical analysis was performed with SPSS (version 22.0, IBM SPSS Inc., Chicago, IL, USA). A p value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 confirmed by a positive polymerase chain reaction test
* Mechanical ventilation

Exclusion Criteria:

* Up to 24 hours on mechanical ventilation
* Severe valvulopathy
* Poor ultrasound window
* Do-not-resuscitate status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe SARS-CoV-2 pneumonia, defined as respiratory failure requiring invasive mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with left ventricle dysfunction (hypokinetic) | 3 month
  Hypokinetic left ventricle function (left ventricle ejection fraction <45%)
Percentage of patients with acute cor pulmonale | 3 month
  Acute cor pulmonale was defined as a dilated right ventricle (right ventricle end-diastolic area/left ventricle end-diastolic area ratio >0.6) associated with the presence of paradoxical septum motion

SECONDARY OUTCOMES:
Differences in respiratory system compliance between patients with and without acute cor pulmonale | Within the first 24 hours of mechanical ventilation.
  Respiratory system compliance is defined as the change in lung volume (Tidal volume, ml) produced by a unit change in pulmonary pressure (driving pressure, cmH2O). The reported value of respiratory system compliance will be reported in ml/cmH2O.
Differences in partial arterial pressure of carbon dioxide (PCO2) between patients with and without acute cor pulmonale | Within the first 24 hours of mechanical ventilation.
  Partial arterial pressure of carbon dioxide will be reported in mmHg.
Differences in PaO2/FiO2 ratio between patients with and without acute cor pulmonale | Within the first 24 hours of mechanical ventilation.
  PaO2/FiO2 ratio is the ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 expressed as a fraction). The reported value is a positive integer.

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816
- [Background] Deng Q, Hu B, Zhang Y, Wang H, Zhou X, Hu W, Cheng Y, Yan J, Ping H, Zhou Q. Suspected myocardial injury in patients with COVID-19: Evidence from front-line clinical observation in Wuhan, China. Int J Cardiol. 2020 Jul 15;311:116-121. doi: 10.1016/j.ijcard.2020.03.087. Epub 2020 Apr 8. PMID 32291207
- [Background] Rath D, Petersen-Uribe A, Avdiu A, Witzel K, Jaeger P, Zdanyte M, Heinzmann D, Tavlaki E, Muller K, Gawaz MP. Impaired cardiac function is associated with mortality in patients with acute COVID-19 infection. Clin Res Cardiol. 2020 Dec;109(12):1491-1499. doi: 10.1007/s00392-020-01683-0. Epub 2020 Jun 14. PMID 32537662
- [Background] Inciardi RM, Lupi L, Zaccone G, Italia L, Raffo M, Tomasoni D, Cani DS, Cerini M, Farina D, Gavazzi E, Maroldi R, Adamo M, Ammirati E, Sinagra G, Lombardi CM, Metra M. Cardiac Involvement in a Patient With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):819-824. doi: 10.1001/jamacardio.2020.1096. PMID 32219357
- [Background] Zeng JH, Liu YX, Yuan J, Wang FX, Wu WB, Li JX, Wang LF, Gao H, Wang Y, Dong CF, Li YJ, Xie XJ, Feng C, Liu L. First case of COVID-19 complicated with fulminant myocarditis: a case report and insights. Infection. 2020 Oct;48(5):773-777. doi: 10.1007/s15010-020-01424-5. Epub 2020 Apr 10. PMID 32277408
- [Background] Szekely Y, Lichter Y, Taieb P, Banai A, Hochstadt A, Merdler I, Gal Oz A, Rothschild E, Baruch G, Peri Y, Arbel Y, Topilsky Y. Spectrum of Cardiac Manifestations in COVID-19: A Systematic Echocardiographic Study. Circulation. 2020 Jul 28;142(4):342-353. doi: 10.1161/CIRCULATIONAHA.120.047971. Epub 2020 May 29. PMID 32469253
- [Background] Dweck MR, Bularga A, Hahn RT, Bing R, Lee KK, Chapman AR, White A, Salvo GD, Sade LE, Pearce K, Newby DE, Popescu BA, Donal E, Cosyns B, Edvardsen T, Mills NL, Haugaa K. Global evaluation of echocardiography in patients with COVID-19. Eur Heart J Cardiovasc Imaging. 2020 Sep 1;21(9):949-958. doi: 10.1093/ehjci/jeaa178. PMID 32556199
- [Background] Mahmoud-Elsayed HM, Moody WE, Bradlow WM, Khan-Kheil AM, Senior J, Hudsmith LE, Steeds RP. Echocardiographic Findings in Patients With COVID-19 Pneumonia. Can J Cardiol. 2020 Aug;36(8):1203-1207. doi: 10.1016/j.cjca.2020.05.030. Epub 2020 May 28. PMID 32474111
- [Background] Helms J, Tacquard C, Severac F, Leonard-Lorant I, Ohana M, Delabranche X, Merdji H, Clere-Jehl R, Schenck M, Fagot Gandet F, Fafi-Kremer S, Castelain V, Schneider F, Grunebaum L, Angles-Cano E, Sattler L, Mertes PM, Meziani F; CRICS TRIGGERSEP Group (Clinical Research in Intensive Care and Sepsis Trial Group for Global Evaluation and Research in Sepsis). High risk of thrombosis in patients with severe SARS-CoV-2 infection: a multicenter prospective cohort study. Intensive Care Med. 2020 Jun;46(6):1089-1098. doi: 10.1007/s00134-020-06062-x. Epub 2020 May 4. PMID 32367170
- [Background] Evrard B, Goudelin M, Montmagnon N, Fedou AL, Lafon T, Vignon P. Cardiovascular phenotypes in ventilated patients with COVID-19 acute respiratory distress syndrome. Crit Care. 2020 May 18;24(1):236. doi: 10.1186/s13054-020-02958-8. No abstract available. PMID 32423461
- [Background] Expert Round Table on Echocardiography in ICU. International consensus statement on training standards for advanced critical care echocardiography. Intensive Care Med. 2014 May;40(5):654-66. doi: 10.1007/s00134-014-3228-5. Epub 2014 Mar 11. No abstract available. PMID 24615559
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Alexandru Popescu B, Waggoner AD; Houston, Texas; Oslo, Norway; Phoenix, Arizona; Nashville, Tennessee; Hamilton, Ontario, Canada; Uppsala, Sweden; Ghent and Liege, Belgium; Cleveland, Ohio; Novara, Italy; Rochester, Minnesota; Bucharest, Romania; and St. Louis, Missouri. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2016 Dec;17(12):1321-1360. doi: 10.1093/ehjci/jew082. Epub 2016 Jul 15. No abstract available. PMID 27422899
- [Background] McLean AS, Needham A, Stewart D, Parkin R. Estimation of cardiac output by noninvasive echocardiographic techniques in the critically ill subject. Anaesth Intensive Care. 1997 Jun;25(3):250-4. doi: 10.1177/0310057X9702500307. PMID 9209605
- [Background] Alam M, Hoglund C, Thorstrand C, Hellekant C. Haemodynamic significance of the atrioventricular plane displacement in patients with coronary artery disease. Eur Heart J. 1992 Feb;13(2):194-200. doi: 10.1093/oxfordjournals.eurheartj.a060146. PMID 1555616
- [Background] Gulati VK, Katz WE, Follansbee WP, Gorcsan J 3rd. Mitral annular descent velocity by tissue Doppler echocardiography as an index of global left ventricular function. Am J Cardiol. 1996 May 1;77(11):979-84. doi: 10.1016/s0002-9149(96)00033-1. PMID 8644649
- [Background] Jardin F, Dubourg O, Bourdarias JP. Echocardiographic pattern of acute cor pulmonale. Chest. 1997 Jan;111(1):209-17. doi: 10.1378/chest.111.1.209. No abstract available. PMID 8996019
- [Background] Mekontso Dessap A, Boissier F, Charron C, Begot E, Repesse X, Legras A, Brun-Buisson C, Vignon P, Vieillard-Baron A. Acute cor pulmonale during protective ventilation for acute respiratory distress syndrome: prevalence, predictors, and clinical impact. Intensive Care Med. 2016 May;42(5):862-870. doi: 10.1007/s00134-015-4141-2. Epub 2015 Dec 9. PMID 26650055
- [Background] Lamia B, Teboul JL, Monnet X, Richard C, Chemla D. Relationship between the tricuspid annular plane systolic excursion and right and left ventricular function in critically ill patients. Intensive Care Med. 2007 Dec;33(12):2143-9. doi: 10.1007/s00134-007-0881-y. Epub 2007 Oct 10. PMID 17928992
- [Background] Edul VS, Ince C, Vazquez AR, Rubatto PN, Espinoza ED, Welsh S, Enrico C, Dubin A. Similar Microcirculatory Alterations in Patients with Normodynamic and Hyperdynamic Septic Shock. Ann Am Thorac Soc. 2016 Feb;13(2):240-7. doi: 10.1513/AnnalsATS.201509-606OC. PMID 26624559